CLINICAL TRIAL: NCT07301112
Title: Transitions and Old Age Potential: Übergänge Und Alternspotenziale (TOP)
Brief Title: Transitions and Old Age Potential - 1st, 2nd, and 3rd Wave
Acronym: TOP
Status: Completed | Type: Observational
Sponsor: Jacobs University Bremen gGmbH (Other)
Collaborators: Federal Institute for Population Research (BIB) (Unknown); German Federal Ministry of the Interior (BMI) (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Sonia Lippke, Head of Health Psychology & Behavioral Medicine Unit, Jacobs University Bremen gGmbH
Other Study IDs: ZA6597V4
Record Dates: First submitted 2025-11-18; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Retirement; Healthy Adults; Elderly
Keywords: longitudinal; cohort study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With the third wave of the Transitions and Old Age Potential (TOP) study, the longitudinal study of initially 5,002 individuals was completed in 2019. Initial findings were published in 2020 through a brochure, policy brief, and methodological report, and presented publicly. The third wave produced two datasets: a panel of 1,561 individuals surveyed across all three waves (2013, 2015/16, 2019) and a couple datasets with 576 complete interviews. Additional data sources such as DEAS, FWS, and SHARE complement the analyses. In 2021, efforts centered on preparing scientific articles for peer-reviewed journals and archiving the third wave at GESIS Leibniz Institute for the Social Sciences, concluding the study that ran from 2011 to 2021.

For further information, see: https://search.gesis.org/research_data/ZA6597 and https://doi.org/10.4232/1.13845

DETAILED DESCRIPTION:
Content and Objectives In 2019, the third wave of the study Transitions and Old Age Potential (TOP) was completed. In addition to the repeated interviews of some of those who had already participated in the study in previous waves, partners were also interviewed. The aim of this supplementary survey was to gain insights into retirement transition in a couple of contexts, focusing on the phenomenon of joint retirement. The initial results were published in June 2020 in the form of a brochure and a policy brief and presented at a press conference. Another publication was the methodological report on the third wave in German and English. In 2021, the focus was on the final editing and submission of the scientific articles from TOP in peer-reviewed journals. The archiving of the third wave of TOP as a scientific use file at GESIS was planned for October 2021. This step concluded the TOP study.

Data and Methods

Within the framework of the third wave of the TOP study, 1,561 persons could be interviewed for the second time. Regarding the partners of these persons, a gross sample of 832 persons resulted, after completion of the last address and panel maintenance of the year 2017/2018. After completion of the field phase of the third wave, 576 complete interviews were available at the couple level. The TOP study thus comprised of two data sets after the completion of the third wave:

the panel data set comprised the persons who had participated in the study on all three survey dates (2013, 2015/2016 and 2019) (1,561 persons) as well as the couple sample with the information provided by the anchors (with current partner from the third survey wave) and the partners from 2019 (576 couple interviews).

In addition to the data from TOP, other studies are also used for the scientific articles, such as the German Ageing Survey (DEAS), the German Volunteer Survey (FWS) and the Survey of Health, Ageing and Retirement in Europe (SHARE).

Duration 01/2011-12/2021

Selected Publications see https://search.gesis.org/research_data/ZA6597

ELIGIBILITY:
Inclusion Criteria:

* aged 55-70
* telephone
* german language

Exclusion Criteria:

* illiterate
* no consent

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The survey is based on a representative sample of 5,002 individuals from the German-speaking residential population, aged between 55 and 70 years (birth cohorts 1942 to 1958). The study focuses on the life plans and potentials of older adults in the labor market, civil society, and family, as well as their transitions into retirement. In spring 2013, a 40-minute telephone interview was conducted using a standardized survey instrument. It included measures in the following areas: sociodemographics, employment and retirement transitions, informal work in civil society and family, perceptions of aging, health and well-being, and personality. In 2015/2016, participants from the first wave who were willing to be re-interviewed were surveyed again. In total, 2,501 interviews were completed at T2
Sampling Method: Probability Sample
Enrollment: 5002 (Actual)
Dates: Start 2013-01-16 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Loneliness | year 2019
  Loneliness was assessed at T3 using three items from the University of California, Los Angeles Loneliness Scale (UCLA-Loneliness Scale) in its short form, based on four-point Likert scales. The loneliness index was calculated as the mean value of the three items with higher means indicating greater loneliness/worse outcome: (0 =never-3=often)
Retirement | years 2013, 2015/2016 and 2019
  Retirement was assessed at T1 by asking participants whether they received a pension or not, with responses transformed into a binary pension/retirement variable (1=yes, 2=no).
Physical Activity (PA) | years 2013, 2015/2016 and 2019
  PA was determined by asking participants how often (<1, 1-2, 3-4, 5+ times per week) they were physically active for more than 30 minutes at T1, T2, and T3.

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Lippke, Principal Investigator — 04212004730

IPD SHARING:
Plan to Share IPD: No
this was not foreseen and consented by data security plan

REFERENCES:
- [Background] https://doi.org/10.4232/1.13845
- See also: study description and further links — https://www.bib.bund.de/EN/Research/Surveys/TOP/transitions-and-old-age-potential.html
- See also: study description and further references — https://search.gesis.org/research_data/ZA6597